CLINICAL TRIAL: NCT00238017
Title: A Randomized, Double Blind Trial on the Efficacy and Safety of Amodiaquine-Artesunate and Amodiaquine Alone in the Treatment of Children With Uncomplicated Falciparum Malaria
Brief Title: Efficacy and Safety of Amodiaquine and Amodiaquine-Artesunate
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: University for Development Studies, Tamale, Ghana (Other); Kintampo Health Research Centre, Ghana (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NP05-M4; A50068
Record Dates: First submitted 2005-10-07; First posted 2005-10-13 (Estimated); Last update posted 2006-02-02 (Estimated); Status verified 2005-07

CONDITIONS: Malaria
Keywords: malaria, amodiaquine, artesunate, safety, efficacy
MeSH Terms: conditions — Malaria

INTERVENTIONS:
Drug: amodiaquine-artesunate versus amodiaquine

SUMMARY:
The purpose of this study is to compare the efficacy and safety of two antimalarial drug regimes, namely amodiaquine versus amodiaquine-artesunate, in the treatment of children with uncomplicated malaria. Also, genetic host factors which might influence efficacy and/or safety will be examined.

DETAILED DESCRIPTION:
Malaria remains a major cause of morbidity and mortality among children in sub-Saharan Africa. Current malaria control largely consists of rapid treatment of patients. Amodiaquine-artesunate and other combinatory treatment regimes including amodiaquine are now being introduced as first-line antimalarial drugs in several African countries. However, data on the efficacy and safety of amodiaquine and amodiaquine-artesunate are scarce. In addition, there is evidence that common genetic host factors, e.g. sickle cell trait, may influence efficacy and safety of these drugs. To examine efficacy and safety of the named drugs as well as a potential influence of genetic host factors on these outcomes a randomized, double blind trial among 400 children with uncomplicated malaria is performed in northern Ghana.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients aged 6 to 59 months
* Body weight >5 kg
* Uncomplicated Plasmodium falciparum malaria
* Mono-infection with P. falciparum with an asexual parasite density between 2,000 to 200,000 parasites/μl
* Axillary temperature ≥37.5°C
* Ability to tolerate oral therapy
* Informed consent by the legal representative of the subject
* Residence in study area

Exclusion Criteria:

* Previous participation in this clinical trial
* Haemoglobin <5 mg/dl
* Mixed plasmodial infection
* Danger signs (unable to drink; repeated vomiting; recent history of convulsions;lethargic or unconscious state; unable to stand up or to sit) and signs of severe malaria as defined by WHO.
* Any other severe underlying disease (cardiac, renal, hepatic diseases, malnutrition, known HIV infection)
* Concomitant disease masking assessment of response
* History of allergy or intolerance against study medications

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400
Dates: Start 2005-10; Study Completion 2005-12

PRIMARY OUTCOMES:
Parasitological and clinical cure rates by days 14 and 28
Parasite and fever clearance times
Carrier rates of sexual parasite stages at days 7, 14 and 28
Incidence rates of adverse events

SECONDARY OUTCOMES:
Incidence rate of haematological and biochemical evidence of drug-induced toxicity
Primary endpoints in children with and without various genetic host factors

CONTACTS AND LOCATIONS:
Overall Officials: Rowland N Otchwemah, PhD, Principal Investigator — University for Development Studies; Frank P Mockenhaupt, MD, Principal Investigator — Malaria Unit, Institute of Tropical Medicine, Charite University, Berlin, Germany; Seth Owusu-Agyei, PhD, Principal Investigator — Kintampo Health Research Centre, Ghana
Locations (1):
- University for Development Studies, Tamale, Northern Region, Ghana